CLINICAL TRIAL: NCT05254379
Title: Transcranial Direct Current Stimulation Treatment for Warriors Experiencing Chronic Pain (tDCS for Warriors)
Brief Title: Transcranial Direct Current Stimulation Treatment for Warriors Experiencing Chronic Pain
Acronym: Warriors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Wounded Warrior Project (Unknown)
Responsible Party: Principal Investigator, Sheila Rauch, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003899
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Post Traumatic Stress Disorder (PTSD); Depression
Keywords: Transcranial direct current stimulation (tDCS); Veterans
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transcranial Direct-Current Stimulation (tDCS) (Experimental): Participants will be assigned to tDCS intervention. Starting Day 1 of EHVP-IOP, remote-based tDCS will be administered with a constant current intensity for 20 min per session for up to 10 sessions over 2 weeks (one session per day) using a Soterix 1x1 tDCS mini-CT Stimulator with headgear and saline-soaked surface sponge electrodes. Therapy sessions will be performed over Zoom. With the exception of day one when the session will occur on its own, the sessions will occur within one hour of the start of the daily therapy session.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — tDCS is a painless brain stimulation treatment that uses direct electrical currents (at a constant, low-intensity level) to stimulate specific parts of the brain and help modulate neuronal activity. Participants will receive a series of tDCS treatments during the Intensive Outpatient Program (IOP) coupled with blood and saliva collections.
  Participants will administer a stimulation session via the Soterix 1x1 tDCS mini-CT Stimulator, after being provided a single-use code to unlock the device by the research staff once proper contact quality is achieved. After the participant enters the unlock code, the screen on the device will show a timer that counts down the minutes until the end of the session. After 20 min, the device will turn off automatically and the study staff will instruct the participant to remove the headset and discard the sponges and to store safely all materials for the next session.

SUMMARY:
The Veteran population has been known to deal with co-morbid chronic pain and PTSD. As a result, they use healthcare services at a higher rate than those Veterans with pain or PTSD alone which leads to an amplified burden on healthcare systems.

tDCS is a painless brain stimulation treatment that uses direct electrical currents (at a constant, low-intensity level) to stimulate specific parts of the brain and help modulate neuronal activity. This study hypothesizes that our short-term therapy-focused treatment program coupled with tDCS administrations will aid in the reduction of chronic pain and PTSD symptoms. Secondly, the investigators intend to examine any relationships between BDNF reduction in reported pain and PTSD and related mental health symptoms. Subjects will be identified from the Emory Healthcare Veterans Program (EHVP-IOP) Veterans and Service members seeking psychiatric treatment for mental health issues including PTSD.

DETAILED DESCRIPTION:
The Veteran population has been known to deal with co-morbid chronic pain and PTSD. As a result, they use healthcare services at a higher rate than those Veterans with pain or PTSD alone which leads to an amplified burden on healthcare systems. In the process of seeking relief and treatment in the healthcare systems, Veterans may use opioid medications to treat chronic pain which puts them at risk for harmful consequences.

This study will be an open trial providing a non-opioid, self-administered, effective pain intervention as part of an effective mental health treatment program. A transcranial direct current stimulation (tDCS) device will be utilized in combination with a cognitive-behavioral therapy (CBT) focused intensive outpatient program (IOP). Additionally, blood and saliva will be collected during this study to perform brain derived neurotropic factor (BDNF) assays comparing outcomes from specific visits: pre-treatment (tx), mid-tx, and post-tx.

The study will take place at the Brain Health Center (BHC) located at 12 Executive Park in the Veterans Program Department.

Subjects will be identified from the Emory Healthcare Veterans Program (EHVP-IOP) Veterans and Service members seeking psychiatric treatment for mental health issues. Incoming patients will be screened for this study and consented prior to the start of their treatment program participation. An electronic consent will be conducted using the REDCap e-Consent framework. A partial waiver of consent is requested to be able to review identifiable information to determine a potential subject's eligibility status.

This study hypothesizes that our short-term therapy-focused treatment program coupled with tDCS administrations will aid in the reduction of chronic pain . Secondly, we intend to examine reductions in PTSD and related mental health symptoms and any relationships between BDNF reduction in reported pain and PTSD and related mental health symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18 -89 years old
* Treated on site for EHVP IOP
* For long-term follow-up, must live in Georgia or Florida
* Eligible for EHVP-IOP PTSD or Unified Protocol tracks
* Willing to self-administer tDCS and complete the measures
* DVPRS pain intensity of 4 or more for most of the day at least 3 days per week
* Have an established PCP (Primary Care Provider) or pain management provider

Exclusion Criteria:

* Implanted pacemaker
* Seizure Disorder
* Pregnancy, if applicable
* Any new onset of the following:

  * Balance problems
  * Difficulty walking
  * Bladder incontinence
  * Bowel incontinence
  * Numbness
  * Tingling
  * Weakness
* Medical contraindications:

  * Current use of sodium channel blockers

    * Lidocaine (OTC/transdermal delivery is ok)
    * Mexiletine
    * Amitriptyline; other tricyclic antidepressants
    * Anti-epileptic medications
* Phenytoin, carbamazepine, lamotrigine, oxcarbazepine, rufinamide, lacosamide and eslicarbazepine acetate

  * Current use of calcium channel blockers
  * Current use of N-Methyl-D-aspartate receptor antagonists

    * Ketamine
    * Dextromethorphan
    * Felbamate
  * History of brain surgery
  * History of brain tumor
  * History of seizure disorder
  * History of stroke
  * Intracranial metal implantation
* Adults unable to consent
* Individuals who are not yet adults
* Prisoners
* Non-English speaking

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Defense and Veterans Pain Rating Scale (DVPRS) | Intake, Days 1,3, 5 and 12 of intervention and at months 1, 3, 6, 9, and 12 of follow-up
  The DVPRS assesses chronic pain using a visual analogue scale of 0 to 10 including general level of pain, and assessment of interference with daily activities, mood, sleep, and stress. It is widely used in clinical care and research and has demonstrated reliability and validity within the military and Veteran population. This is a clinical measure collected per standard of care at intake. However, this measure will be collected for research purposes at additional timepoints, include each tDCS session, 1-10, and all follow-up visits.

SECONDARY OUTCOMES:
Changes in PROMIS 3a pain intensity | Day 1 and 12 of intervention and at months 1, 3, 6, 9, and 12 of follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pain 3a Intensity instrument assesses how much a person hurts via the following 3 questions rated on a 1 (no pain) to 5 (very severe) point scale: "In the past 7 days: How intense was your pain at its worst? How intense was your average pain? What is your level of pain right now?" Per the PROMIS measure website, "The Pain Intensity short form is universal rather than disease- specific. The first two items within the short form assess pain intensity over the past seven days while the last item asks patient to rate their pain intensity 'right now'." This is a research-specific measure collected for enrolled participants only and will take approximately 10 minutes to complete.
  Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function.
Changes in PROMIS 8a pain interference | Day 1 and 12 of intervention and at months 1, 3, 6, 9, and 12 of follow-up
  The PROMIS Pain Interference instrument measures the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities via 8 items. Pain Interference also incorporates items probing sleep and enjoyment in life, though the item bank only contains one sleep item. The Pain Interference short form is universal rather than disease-specific. The Pain Interference items utilize a 7-day recall period (items include the phrase "the past 7 days").
  Items are rated on a 1 (not at all) to 5 (very much) point scale, such as the following questions: In the past 7 days, "How much did pain interfere with your day-to-day activities?" "How much did pain interfere with the things you usually do for fun?" etc.
Changes in PTSD Checklist- PCL-5 | Days 1 through 12 of intervention and at months 1, 3, 6, 9, and 12 of follow-up
  The PCL-5 is a 20-item self-report measure of PTSD severity in the past month with 4 subscales: Intrusion symptoms (items 1- 5); Avoidance symptoms (items 6-7); negative cognitions and mood symptoms (items 8-14) and Hyperarousal symptoms (items 15-20). Each item ranges from 0 (not at all) to 4 (extremely). Cut points and psychometrics are pulled from the most recent studies on the new PCL-5. This is a clinical measure collected per standard of care.
Changes in BDNF in saliva | Days 2, 5 and 11 of the intervention
  Collection of saliva will be done pre tDCS, prior to the Therapy Session, and post-Therapy Session. Saliva will be assayed to examine Brain-derived neurotrophic factor (BDNF) and change in BDNF over the intervention session.
  The study team will collect these samples from all participants to test feasibility and reliability of saliva as a clinically useful BDNF source.
Changes in BDNF in blood | Days 2, 5 and 11 of the intervention
  Collection of blood will be done pre tDCS, prior to the Therapy Session, and post-Therapy Session. Blood will be assayed to examine Brain-derived neurotrophic factor (BDNF) and change in BDNF over the intervention session.
PTSD Checklist - Stressor-Specific Version (PCL-5 | Intake, Days 1,3, 5 and 12 of intervention and at months 1, 3, 6, 9, and 12 of follow-up
  The PCL-5 is a 20-item self-report measure of PTSD severity in the past month with 4 subscales: Intrusion symptoms (items 1- 5); Avoidance symptoms (items 6-7); negative cognitions and mood symptoms (items 8-14) and Hyperarousal symptoms (items 15-20). Each item ranges from 0 (not at all) to 4 (extremely). Cut points and psychometrics are pulled from the most recent studies on the new PCL-5.
Patient Health Questionnaire- 9 (PHQ-9) | Intake, Days 1,3, 5 and 12 of intervention
  The PHQ-9 is a 9 item, well-validated measure of depression and secondary outcome. The PHQ-9 assesses symptoms of major depression in the past two weeks from 0 (not at all) to 3 (nearly every day) and has excellent internal and test-retest reliability as well as construct and criterion validity (80). The PHQ-9 is effective in detecting treatment changes in depression in PC settings.
Change in Clinician Administered PTSD Scale-5 (CAPS5) | Intake, Day 1 of treatment and month 3 follow up
  CAPS is an interview measure of PTSD severity that is collected for the purposes of the clinical treatment program (standard of care). Current PTSD will be assessed by assessors in relation to the trauma that is currently most upsetting. The CAPS-5 has excellent psychometrics and requires about 45 minutes to complete. 20% of CAPS will be rated by a second rater to ensure reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Rauch, PhD, Principal Investigator — Emory University; Barbara O Rothbaum, Principal Investigator — Emory University; Boadie W Dunlop, MD, Principal Investigator — Emory University
Locations (1):
- Emory Division of Psychiatry, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT05254379/ICF_001.pdf